CLINICAL TRIAL: NCT03385824
Title: Self-Advocacy for Independent Life (SAIL) After Traumatic Brain Injury
Brief Title: Self-Advocacy for Independent Life (SAIL) After TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Lenore Hawley, Principal Investigator, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NIDILRR SAIL 2017
Record Dates: First submitted 2017-12-19; First posted 2017-12-29 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: traumatic brain injury; advocacy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Advocacy for Independent Life (SAIL) (Experimental): 10 week treatment program to improve self-advocacy skills. Includes 4 in-person group sessions (3 hours per session) and two supportive phone calls; workbook and home assignments.
  Interventions: Behavioral: Self-Advocacy for Independent Life (SAIL)
- Control (No Intervention): SAIL workbook provided at the conclusion of the study.

INTERVENTIONS:
Behavioral: Self-Advocacy for Independent Life (SAIL) — SAIL program is based on an interactive workshop model. In -person sessions will focus on: enhancement of self-efficacy beliefs; enhancement of knowledge of TBI self-advocacy information; group process to instill hope and universality; and practice of self-advocacy behaviors in a supportive neuro-rehabilitation structured group environment.
  Arms: Self-Advocacy for Independent Life (SAIL)

SUMMARY:
Traumatic brain injury (TBI) has been conceptualized as a chronic health condition, warranting self-advocacy for health management services across the lifespan. Successful self-advocacy requires a combination of cognitive and communication skills (problem solving, organization, negotiation, etc), which may be impaired following TBI. This project focuses on developing and testing the efficacy of an intervention to enhance self-advocacy skills in individuals who have sustained TBI. This two-arm, randomized controlled trial will include approximately 74 participants, recruited in 4 waves of approximately 18-20 per wave, with each wave recruited from a different geographic area of the state. The primary hypothesis states that participants receiving the treatment intervention will demonstrate significantly greater improvements in self-advocacy beliefs (SAS) from baseline to post-intervention as compared to participants in the control group. Treatment will consist of interactive 4-session workshops along with 2 booster phone calls. Control participants will receive a copy of a self-advocacy workbook after all assessments are completed. Baseline, post-treatment and two follow-up assessments will take place.

ELIGIBILITY:
Inclusion Criteria:

* Documented TBI due to an external mechanical force
* Received inpatient or outpatient rehabilitation for TBI
* At least 9 months post TBI
* Able to travel independently in the community
* Able to attend intervention sessions

Exclusion Criteria:

* Unable to read or speak English well enouth to complete assessments and actively participate in study intervention
* Currently in inpatient TBI rehabilitation
* Previously participated in a SAIL program
* Participating in another research trial
* Unable to perform neuropsychological baseline assessment
* Score of 30 or above on GSES

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Self-Advocacy Scale (SAS) | Change in SAS score from Baseline to 11 weeks (immediately post-tx)
  The Self-Advocacy Scale (SAS) is an eight-item 1-4 Likert rating scale (1 = not confident to 4 = very confident), conceptualized as a domain specific self-efficacy scale. The SAS is designed to measure an individual's current beliefs about his or her ability to produce desired self-advocacy outcomes. Scores range from 8 to 32 with higher scores indicative of better self-advocacy skills.
Self-Advocacy Scale (SAS) | Change in SAS score from Baseline to 17 weeks (6 weeks post-tx)
  The Self-Advocacy Scale (SAS) is an eight-item 1-4 Likert rating scale (1 = not confident to 4 = very confident), conceptualized as a domain specific self-efficacy scale. The SAS is designed to measure an individual's current beliefs about his or her ability to produce desired self-advocacy outcomes. Scores range from 8 to 32 with higher scores indicative of better self-advocacy skills.
Self-Advocacy Scale (SAS) | Change in SAS score from Baseline to 23 weeks (12 weeks post-tx)
  The Self-Advocacy Scale (SAS) is an eight-item 1-4 Likert rating scale (1 = not confident to 4 = very confident), conceptualized as a domain specific self-efficacy scale. The SAS is designed to measure an individual's current beliefs about his or her ability to produce desired self-advocacy outcomes. Scores range from 8 to 32 with higher scores indicative of better self-advocacy skills.

SECONDARY OUTCOMES:
Personal Advocacy Activity Scale (PAAS) | Change in PAAS score from Baseline to 11 weeks (immediately post-tx)
  The Personal Advocacy Activity Scale (PAAS) is a 12-item self-rating of personal advocacy behaviors. Participants respond to each item by indicating how frequently they perform each activity, "Not at all", "1 - 4 times", or "5 or more times". Scores range from 12 to 36 with higher scores indicating more personal advocacy behavior.
Personal Advocacy Activity Scale (PAAS) | Change in PAAS score from Baseline to 17 weeks (6 weeks post-tx)
  The Personal Advocacy Activity Scale (PAAS) is a 12-item self-rating of personal advocacy behaviors. Participants respond to each item by indicating how frequently they perform each activity, "Not at all", "1 - 4 times", or "5 or more times". Scores range from 12 to 36 with higher scores indicating more personal advocacy behavior.
Personal Advocacy Activity Scale (PAAS) | Change in PAAS score from Baseline to 23 weeks (12 weeks post-tx)
  The Personal Advocacy Activity Scale (PAAS) is a 12-item self-rating of personal advocacy behaviors. Participants respond to each item by indicating how frequently they perform each activity, "Not at all", "1 - 4 times", or "5 or more times". Scores range from 12 to 36 with higher scores indicating more personal advocacy behavior.
General Self Efficacy Scale (GSES) | Change in GSES score from Baseline to 11 weeks (immediately post-tx)
  General Self Efficacy Scale (GSES) is a 10-item Likert rating scale assessing beliefs about one's ability to cope with various demands in life, a core component of self-advocacy.The GSES produces a single score ranging from 10 to 40, with higher scores indicating greater general self-efficacy.
General Self Efficacy Scale (GSES) | Change in GSES score from Baseline to 17 weeks (6 weeks post-tx)
  General Self Efficacy Scale (GSES) is a 10-item Likert rating scale assessing beliefs about one's ability to cope with various demands in life, a core component of self-advocacy.The GSES produces a single score ranging from 10 to 40, with higher scores indicating greater general self-efficacy.
General Self Efficacy Scale (GSES) | Change in GSES score from Baseline to 23 weeks (12 weeks post-tx)
  General Self Efficacy Scale (GSES) is a 10-item Likert rating scale assessing beliefs about one's ability to cope with various demands in life, a core component of self-advocacy.The GSES produces a single score ranging from 10 to 40, with higher scores indicating greater general self-efficacy.
Satisfaction With Life Scale (SWLS) | Change in SWLS score from Baseline to 11 weeks (immediately post-tx)
  The Satisfaction with Life Scale (SWLS) is a subjective, five-item 1-7 Likert rating scale measuring global life satisfaction - a cognitive self-assessment of quality of life. Scores range from 5 to 35 with higher scores indicative of greater life satisfaction
Satisfaction With Life Scale (SWLS) | Change in SWLS score from Baseline to 17 weeks (6 weeks post-tx)
  The Satisfaction with Life Scale (SWLS) is a subjective, five-item 1-7 Likert rating scale measuring global life satisfaction - a cognitive self-assessment of quality of life. Scores range from 5 to 35 with higher scores indicative of greater life satisfaction
Satisfaction With Life Scale (SWLS) | Change in SWLS score from Baseline to 23 weeks (12 weeks post-tx)
  The Satisfaction with Life Scale (SWLS) is a subjective, five-item 1-7 Likert rating scale measuring global life satisfaction - a cognitive self-assessment of quality of life. Scores range from 5 to 35 with higher scores indicative of greater life satisfaction
Flourishing Scale (FS) | Change in total Flourishing Scale score from Baseline to 11 weeks (immediately post-tx)
  The Flourishing Scale (FS) is a brief eight-item, self-rated, 1-7 point Likert scale measure of self-perceived success in areas such as social relationships, self-esteem, and purpose in life. Scores range from 5 to 35 with higher scores indicating better self-perceived success.
Flourishing Scale (FS) | Change in total Flourishing Scale from Baseline to 17 weeks (6 weeks post-tx)
  The Flourishing Scale (FS) is a brief eight-item, self-rated, 1-7 point Likert scale measure of self-perceived success in areas such as social relationships, self-esteem, and purpose in life. Scores range from 5 to 35 with higher scores indicating better self-perceived success.
Flourishing Scale (FS) | Change in total Flourishing Scale score from Baseline to 23 weeks (12 weeks post-tx)
  The Flourishing Scale (FS) is a brief eight-item, self-rated, 1-7 point Likert scale measure of self-perceived success in areas such as social relationships, self-esteem, and purpose in life. Scores range from 5 to 35 with higher scores indicating better self-perceived success.
Participation Assessment with Recombined Tools-Objective (PART-O) | Change in PART-O score from Baseline to 11 weeks (immediately post-tx)
  Objective measure of participation in society
Participation Assessment with Recombined Tools-Objective (PART-O) | Change in PART-O score from Baseline to 17 weeks (6 weeks post-tx)
  Objective measure of participation in society
Participation Assessment with Recombined Tools-Objective (PART-O) | Change in PART-O score from Baseline to 23 weeks (12 weeks post-tx)
  Objective measure of participation in society

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No